CLINICAL TRIAL: NCT00410475
Title: Cancer Risk in X-Ray Technologists
Brief Title: Cancer Risk in X-Ray Technologists: Second Survey
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999997053; OH97-C-N053
Record Dates: First submitted 2006-12-12; First posted 2006-12-13 (Estimated); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Radiation-Induced Neoplasms; Breast+Neoplasm+Radiation+Etiology; Thyroid+Neoplasm+Radiation+Etiology
Keywords: Ionizing Radiation; Cohort Study; Radiation-Induced Neoplasms; Radiologic Technologists; Ultraviolet Radiation
MeSH Terms: conditions — Neoplasms, Radiation-Induced

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- U.S. radiologic technologists: Radiologic technologists certified by the American Registry of Radiologic Technologists (ARRT) during 1923-1980 and residing in any U.S. state or territory.

SUMMARY:
Researchers at the National Cancer Institute and the University of Minnesota have followed a nationwide cohort of 146,022 radiologic technologists since 1982 (Boice 1992; Doody 1998; Mohan 2003; Sigurdson 2003). This is one of the largest cohorts of medical radiation workers studied to date (Yoshinaga 2003)and the only one with substantial numbers of women (73% female), extensive covariate data, both incident and death outcomes, and estimated occupational radiation doses. The overall study objectives are to: quantify radiation dose-response for cancers of the breast, thyroid, and other radiogenic sites; assess cancer risks associated with genotypic, phenotypic, or other biologically measurable factors; and determine if genetic variation modifies radiation-related cancer risks.

More than 110,000 technologists completed at least one of three comprehensive questionnaire surveys administered over the last 20 years and 18,500 are deceased. The First Survey was mailed during 1984-1989 to 132,454 known living radiologic technologists, of whom 90,305 (68%) completed the survey (Boice 1992). The Second Survey was mailed during 1993-1998 to 126,628 known living technologists, of whom 90,972 (72%) completed the questionnaire (Sigurdson2003). Both surveys included detailed questions about employment as a radiologic technologist, family history of cancer, reproductive history, height, weight, other cancer risk factors (such as alcohol and tobacco use), history of personal diagnostic and therapeutic medical radiation procedures, and information on cancer and other health outcomes. A third follow-up of this cohort was recently completed. During 2003-2005, the Third Survey was mailed or administered by telephone to 101,694 living cohort members who had completed at least one of the two previous surveys; 73,838 technologists (73%) completed the survey. This questionnaire elicited information on medical outcomes to assess radiation-related risks, detailed calendar-specific employment data to refine the occupational ionizing radiation dose estimates, and behavioral and residential histories for estimating lifetime ultraviolet (UV) radiation exposures.

The large number of women with estimates of cumulative radiation dose to specific organs (e.g. breast) (Simon 2006; see Figure 7 and Table 9) offers at are opportunity to study effects of low-dose radiation exposure on breast and thyroid cancers, the two most sensitive organ sites for radiation carcinogenesis in women.. We are not aware of any other study population in which both quantified radiation doses and biospecimens are available for individuals with protracted low-dose ionizing radiation exposures. Incorporation of assessment of the role of genetic polymorphisms and molecular variants in DNA repair and other genetic pathways that may be functionally important in radiation carcinogenesis would provide initial results on the possible role of genetic factors in the cancer-radiation relationship. Because large numbers of women are exposed to ubiquitous low-dose radiation from occupational, medical, and environmental sources, the presence of radiation-sensitive genetic variants that influence the risk of breast and other cancers would have important public health implications.

DETAILED DESCRIPTION:
BACKGROUND:

The Radiation Epidemiology Branch and the University of Minnesota have followed a nationwide cohort of 146,022 U.S. radiologic technologists (USRT) since 1982 to assess cancer and other disease risks associated with long-term repeated low doses of ionizing radiation. The USRT Study is the largest cohort of medical radiation workers studied to date and the only one with substantial numbers of women, extensive covariate data, incident and fatal cancer and other outcomes, estimates of individual historical occupational radiation doses, personal medical radiation doses, and personal and residential solar ultraviolet radiation (UVR) doses, and biospecimens for breast and thyroid cancer cases and comparison subjects. This cohort is uniquely suited for addressing outstanding scientific questions about differences in risk related to the nature of radiation exposure, specifically whether risks are the same from a single or a few high-dose exposures (e.g. atomic bomb, radiotherapy) or from many small exposures over time that might be mitigated by DNA repair or other mechanisms. The nationwide distribution of the cohort, with wide-ranging UVR exposures, also offers a rare opportunity to evaluate risks for non-melanoma skin cancer with UVR, which will be a major focus of study during the next few years.

OBJECTIVES:

1. Assess risks of cancer and other diseases from long-term low-dose occupational and personal medical exposures.
2. Assess risks of cancer and other diseases from occupational exposure to emerging and evolving radiologic modalities (i.e. nuclear medicine, fluoroscopically-guided procedures).
3. Assess risks of skin and other cancers from solar ultraviolet radiation exposures.
4. Conduct discovery of genetic determinants for thyroid cancer and rapid replication of main genotype effects for breast cancer.
5. Evaluate gene-radiation and ionizing radiation-ultraviolet radiation interactions.

ELIGIBILITY:

All radiologic technologists certified by the American Registry of Radiologic Technologists for at least two years during 1926-1982 were eligible for study. Excluded were technologists who resided outside the U.S.

DESIGN:

Cohort study: The full USRT cohort consists of 146,022 radiologic technologists. The cohort is predominantly female (73%), Caucasian (93%), and presently 67 years old on average; 83% are living and 16% are deceased or presumed deceased. Three questionnaire surveys were conducted during 1983-2005 to collect information on occupational, personal medical, and personal and ambient residential ultraviolet radiation exposures, other cancer risk factors, and cancer and other disease outcomes. More than 110,000 technologists participated in the first and/or second surveys. The most recent follow-up (third survey) was conducted during 2003-2005 to obtain detailed work history information for improving occupational dosimetry. Enhanced estimates of individual annual badge dose (personal dose equivalent) and radiation absorbed doses to 12 organs and tissues (breast, thyroid, brain, red bone-marrow, lung, heart, ovary, colon, testes, skin of extremities, skin of head and neck, and lens of eye) were recently completed for survey participants. Linear dose-response analyses are underway to quantify risks from protracted low-dose radiation for cancers (e.g., breast, thyroid) and other radiation-related diseases (e.g., cardiovascular, cataracts). A fourth questionnaire survey is under development and will collect information on cancer and other disease outcomes, work history with nuclear medicine and fluoroscopically-guided procedures, and other risk factors. Fourth survey outcomes will be used to assess incident cancer risks with UVR exposure data collected on the third survey. Collection of blood or buccal cell samples from breast and thyroid cancer cases and comparison subjects continues. Future plans include a case-control study of basal cell carcinoma to assess risks with ultraviolet and ionizing radiation exposure, genetic variants, and interactions.

ELIGIBILITY:
* INCLUSION CRITERIA:

Medical x-ray technologists certified (at least two years during 1926-1982) by the American Registry of Radiologic Technicians (ARRT).

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible radiologic technologists certified by ARRT
Sampling Method: Probability Sample
Enrollment: 146022 (Actual)
Dates: Start 1997-09-17 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Ionizing radiation | Work history information collected on questionnaires plus badge dose measurements
  Occupational ionizing radiation-related risks for cancer and other medical outcomes.

SECONDARY OUTCOMES:
Ultraviolet radiation | Sun exposure information and medical outcomes
  Cancer and other disease risks associated with ultraviolet radiation exposure.

CONTACTS AND LOCATIONS:
Overall Officials: Cari M Kitahara, Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] Simon SL, Preston DL, Linet MS, Miller JS, Sigurdson AJ, Alexander BH, Kwon D, Yoder RC, Bhatti P, Little MP, Rajaraman P, Melo D, Drozdovitch V, Weinstock RM, Doody MM. Radiation organ doses received in a nationwide cohort of U.S. radiologic technologists: methods and findings. Radiat Res. 2014 Nov;182(5):507-28. doi: 10.1667/RR13542.1. Epub 2014 Oct 31. PMID 25361400
- [Background] Preston DL, Kitahara CM, Freedman DM, Sigurdson AJ, Simon SL, Little MP, Cahoon EK, Rajaraman P, Miller JS, Alexander BH, Doody MM, Linet MS. Breast cancer risk and protracted low-to-moderate dose occupational radiation exposure in the US Radiologic Technologists Cohort, 1983-2008. Br J Cancer. 2016 Oct 25;115(9):1105-1112. doi: 10.1038/bjc.2016.292. Epub 2016 Sep 13. PMID 27623235
- [Background] Kitahara CM, Preston DL, Neta G, Little MP, Doody MM, Simon SL, Sigurdson AJ, Alexander BH, Linet MS. Occupational radiation exposure and thyroid cancer incidence in a cohort of U.S. radiologic technologists, 1983-2013. Int J Cancer. 2018 Nov 1;143(9):2145-2149. doi: 10.1002/ijc.31270. Epub 2018 Feb 2. PMID 29355960